CLINICAL TRIAL: NCT06828744
Title: Effectiveness of Dorsal Glide Mobilization of the Ankle Joint on Range of Motion and Performance in Young Basketball Athletes With Unilateral Restricted Ankle Dorsiflexion: A Randomized Controlled Trial
Brief Title: Effectiveness of Dorsal Glide Mobilization on Ankle Mobility and Basketball Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: International Hellenic University (Other)
Responsible Party: Principal Investigator, Dimitrios Lytras, Dimitrios Lytras, Assistant Professor in the Department of Physiotherapy at the International Hellenic University, International Hellenic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EC-2/2025
Record Dates: First submitted 2025-02-11; First posted 2025-02-14 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Unilateral Restricted Ankle Dorsiflexion
Keywords: Unilateral Restricted Ankle Dorsiflexion; Range of motion (ROM); Eccentric exercise; Posterior talocrural glide; Basketball athletes
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial will be conducted, including 38 young basketball athletes with confirmed restricted ankle dorsiflexion ROM. Participants will be randomly assigned to an intervention group and a control group. Both groups will follow a five-week training program consisting of eccentric exercises and stretching, performed two times per week, to improve athletic performance. The intervention group, in addition to the exercise program, will undergo ankle joint mobilization sessions for the same duration.
Who Masked: Outcomes Assessor
Masking Description: A masked assessor will conduct the measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Group (Active Comparator): Participants will follow an exercise and stretching program for five weeks, performed two times per week.
  The program will consist of eccentric strengthening and stretching exercises targeting the gastrocnemius and soleus muscles. The eccentric strengthening component will include heel-lowering exercises. For the gastrocnemius, the participant will stand on an elevated surface with the knee fully extended and will slowly lower the heel. For the soleus, the participant will perform the same movement with the knee slightly flexed. Participants will perform three sets of fifteen repetitions for each exercise, with approximately one-minute rest intervals between sets. In addition, step-lunge dorsiflexion drills will be performed to promote functional dorsiflexion under load.
  The stretching component will focus on the gastrocnemius and soleus muscles. The gastrocnemius stretch will be performed in a lunge position with both heels on the ground and the back knee extended, while the soleus
  Interventions: Other: Exercise
- Exercise + Joint mobilization (Experimental): In addition to the exercise and stretching program followed by the control group, participants will receive a manual therapy program targeting talocrural joint arthrokinematics, delivered twice per week for five weeks by the same physiotherapist. Each supervised session will last approximately 25 minutes.
  The manual therapy protocol will include posterior talar glide mobilization with active dorsiflexion according to the mobilization-with-movement concept. This technique will be applied for three sets of ten repetitions using grade III-IV oscillatory mobilizations. In addition, posterior talar glide mobilizations will be applied in non-weight-bearing conditions, as well as in weight-bearing using a stabilization belt, while the participant actively dorsiflexes the ankle within a pain-free range.
  Furthermore, participants will be instructed to perform a talocrural joint self-mobilization technique using a belt at home, performed daily for three sets of 30 to 60 seconds.
  Interventions: Other: Exercise plus Joint Mobilization

INTERVENTIONS:
Other: Exercise — Participants in this group will follow an exercise and stretching program for five weeks, performed two times per week.
  Arms: Exercise Group
Other: Exercise plus Joint Mobilization — Participants in this group will follow a five-week exercise and stretching program, performed two times per week, in combination with an ankle joint mobilization program.
  Arms: Exercise + Joint mobilization

SUMMARY:
Background: Ankle dorsiflexion is a crucial factor for functional lower limb performance, particularly in sports like basketball, where dynamic movements, direction changes, jumps, and landings are essential for athletic success. Eccentric exercise has been shown to improve dorsiflexion range of motion (ROM), enhancing muscle strength, flexibility, and athletic performance. Additionally, ankle joint mobilization, specifically posterior talocrural glide, has demonstrated promising results in improving mobility, restoring ROM, and reducing compensatory movement strategies. However, the combined effects of eccentric exercise and joint mobilization on increasing ankle dorsiflexion ROM and improving athletic performance in young basketball athletes have not yet been sufficiently investigated.

Objective: The purpose of this study is to investigate the effectiveness of combining eccentric exercise and posterior talocrural glide mobilization in improving ankle dorsiflexion ROM and enhancing athletic performance in young basketball athletes.

Methods: A randomized controlled trial will be conducted, including 38 young basketball athletes with confirmed restricted ankle dorsiflexion ROM. Participants will be randomly assigned to an intervention group and a control group. Both groups will follow a five-week training program consisting of eccentric exercises and stretching, performed two times per week, to improve athletic performance. The intervention group, in addition to the exercise program, will undergo ankle joint mobilization sessions for the same duration.

Ankle dorsiflexion ROM, maximum isometric strength of the ankle muscles, fatigue resistance through specific endurance tests, and performance via functional tests will be assessed at baseline, at the end of the five-week program, and three months after the intervention. Statistical analysis will be conducted using a two-way repeated-measures ANOVA, with the significance level set at p < 0.05.

DETAILED DESCRIPTION:
Background: Ankle dorsiflexion is a crucial factor for functional lower limb performance, particularly in sports like basketball, where dynamic movements, direction changes, jumps, and landings are essential for athletic success. Eccentric exercise has been shown to improve dorsiflexion range of motion (ROM), enhancing muscle strength, flexibility, and athletic performance. Additionally, ankle joint mobilization, specifically posterior talocrural glide, has demonstrated promising results in improving mobility, restoring ROM, and reducing compensatory movement strategies. However, the combined effects of eccentric exercise and joint mobilization on increasing ankle dorsiflexion ROM and improving athletic performance in young basketball athletes have not yet been sufficiently investigated.

Objective: The purpose of this study is to investigate the effectiveness of combining eccentric exercise and posterior talocrural glide mobilization in improving ankle dorsiflexion ROM and enhancing athletic performance in young basketball athletes.

Methods: A randomized controlled trial will be conducted, including a total of 38 young basketball athletes with confirmed restricted ankle dorsiflexion ROM. Participants will be randomly assigned to an intervention group and a control group. Both groups will follow a five-week training program consisting of eccentric exercises and stretching, performed two times per week, to improve athletic performance. In addition, all participants will continue their regular basketball-specific and plyometric team training throughout the study period, ensuring equivalent overall training exposure between groups and controlling for potential confounding effects of training load. The intervention group, in addition to the exercise program, will undergo ankle joint mobilization sessions for the same duration, whereas the control group will not receive joint mobilization.

Ankle dorsiflexion ROM, maximum isometric strength of the ankle muscles, fatigue resistance through specific endurance tests, and performance via functional tests will be assessed at baseline, at the end of the five-week program, and three months after the intervention. Statistical analysis will be conducted using a two-way repeated-measures ANOVA, with the significance level set at p < 0.05.

Expected Outcomes: Improvements in ankle dorsiflexion ROM, muscle strength, and athletic performance are expected, along with a reduction in fatigue and compensatory movement strategies. The intervention is also anticipated to enhance ankle stability and lower the risk of injuries.

ELIGIBILITY:
Inclusion Criteria:

* Participants healthy and actively engaged in basketball training at the time of the study.
* No presence of ankle pain or use of medication for musculoskeletal injuries or pain management at the time of the study.
* Participation in regular training for at least one month prior to the study.
* A restriction in ankle dorsiflexion of at least 2 cm in one foot compared to the other, as measured using the Weight-Bearing Lunge Test (WBLT).
* Written informed consent must be provided before participation in the study.

Exclusion Criteria:

* History of lower extremity surgery.
* Musculoskeletal injury to the lower extremity within the past six months.
* Presence of neurological, vestibular, or balance disorders, or diagnosed connective tissue disease.
* Inability to comply with the intervention or assessment procedures.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-11-30 (Actual); Study Completion 2025-11-30 (Actual)

PRIMARY OUTCOMES:
Active Range of Motion of Ankle Dorsiflexion using a Digital Goniometer | Baseline, end of 5th week, 3-moth follow-up
  The active range of motion (ROM) of ankle dorsiflexion will be measured using a digital goniometer, which provides joint angle measurements. The measurement will be performed with the participant in a seated position and the knee slightly flexed. The goniometer will be placed on the lateral malleolus and aligned with the axis of the tibia and the foot. The athlete will perform maximum active dorsiflexion, and the angle (in degrees) formed between the tibia and the foot will be recorded. Three trials will be performed and the mean value will be used for analysis. This measurement provides information regarding ankle mobility and helps identify potential motion restrictions. The use of a digital goniometer for ROM assessment is widely applied in clinical and research settings when standardized procedures are followed.
Dorsiflexion Range of Motion in a Closed Kinetic Chain using the Weight-Bearing Lunge Test (WBLT) | Baseline, end of 5th week, 3-moth follow-up
  The Weight-Bearing Lunge Test (WBLT) is used to assess the range of motion (ROM) of ankle dorsiflexion in a closed kinetic chain. The test is performed with the participant standing facing a wall and advancing the tibia while keeping the heel in contact with the ground. The toe-to-wall distance (in cm) is measured while the knee remains in contact with the wall. Three trials are recorded and the mean value is used for analysis. This test provides a functional measure of ankle dorsiflexion under weight-bearing conditions and is widely used in both clinical and research settings.

SECONDARY OUTCOMES:
Maximum Isometric Strength of Ankle Dorsiflexors and Plantar Flexors using a Handheld Dynamometer | Baseline, end of 5th week, 3-moth follow-up
  The maximum isometric strength of the ankle dorsiflexors and plantar flexors will be assessed using a handheld dynamometer. Measurements will be performed with the participant in a seated position, with the hip and knee at approximately 90° and the ankle in a neutral position. The device will be applied to the foot while the athlete performs a maximal voluntary isometric contraction in both dorsiflexion and plantarflexion. Three maximal contractions will be recorded for each muscle group, and the highest value of force output (in Newtons, N) will be used for analysis. This method provides information regarding ankle muscle strength and functional capacity and is widely used in clinical and research settings when standardized procedures are applied.
Jump Height (cm) using the Countermovement Jump (CMJ) Test | Baseline, end of 5th week, 3-moth follow-up
  The Countermovement Jump (CMJ) test is used to assess the explosive power of the lower limb muscles. Jump height (in cm) will be recorded using an optical measurement system, which calculates jump height based on flight time. Participants will perform one familiarization trial followed by three valid jumps, and the mean value will be used for analysis. This test provides an indicator of lower-limb explosive power and neuromuscular performance and is widely used in athletic populations.
Endurance and Fatigue Resistance using the Fatigue Index (FI) derived from repeated single-leg hops | Baseline, end of 5th week, 3-moth follow-up
  The Fatigue Index (FI) is used to assess lower-limb fatigue resistance during repeated single-leg hopping. The FI is calculated as the relative change in performance between the initial and the final phase of repeated hop efforts, with higher values indicating a greater decline in performance. This measure provides information about the athlete's ability to maintain functional performance under repeated loading conditions and complements absolute performance measures obtained from hop tests.
Performance Assessment using the Single-Leg 6m Timed Hop Test | Baseline, end of 5th week, 3-moth follow-up
  The Single-Leg 6 m Timed Hop Test is used to evaluate speed, explosive power, and balance control during repeated hopping movements. The athlete performs consecutive single-leg hops over a total distance of 6 meters. The time (in seconds) is recorded using a stopwatch, starting when the athlete's heel lifts from the ground in the initial position and stopping when the test foot crosses the finish line. The time is measured to the nearest tenth of a second. The athlete performs one familiarization trial followed by two valid trials, and the mean value of the two trials is used for analysis.
Performance Assessment using the Triple Hop for Distance Test | Baseline, end of 5th week, 3-moth follow-up
  The Triple Hop for Distance Test is used to evaluate explosive power, balance control, and dynamic ankle stability. The athlete stands on one leg and performs three consecutive forward hops, always landing on the same foot while maintaining balance. The total hop distance (in centimeters) is measured from the starting position to the final landing point using a measuring tape placed on the ground. The athlete performs one familiarization trial followed by two valid trials, and the mean value of the two trials is used for analysis.
Performance Assessment using the Single-Leg Hop Test for Distance | Baseline, end of 5th week, 3-moth follow-up
  The Single-Leg Hop Test for Distance is used to assess explosive power, balance, and ankle joint stability. The athlete stands on the test leg, performs a maximal forward jump, and lands on the same foot while attempting to maintain balance. The jump distance (in centimeters) is measured from the starting position to the landing point with a measuring tape placed on the ground. The athlete performs one familiarization trial followed by two valid trials, and the mean value of the two trials is used for analysis.
Strength Endurance and Explosiveness assessed using the Reactive Strength Index (RSI) | Baseline, end of 5th week, 3-moth follow-up
  The Reactive Strength Index (RSI) is used to evaluate an athlete's ability to rapidly transition from eccentric to concentric muscle action during stretch-shortening cycle activities. Participants will perform repeated jump contacts with minimal ground contact time. RSI will be calculated as jump height divided by ground contact time, and the mean value of valid trials will be used for analysis. This assessment provides an indicator of reactive and explosive neuromuscular performance.

CONTACTS AND LOCATIONS:
Locations (1):
- International Hellenic University, Thessaloniki, Greece, Greece

IPD SHARING:
Plan to Share IPD: No